CLINICAL TRIAL: NCT04254874
Title: An Open, Prospective/Retrospective, Randomized Controlled Cohort Study to Compare the Efficacy of Two Therapeutic Schemes(Abidol Hydrochloride,Abidol Hydrochloride Combined With Interferon Atomization)in the Treatment of 2019-nCoV Pneumonia.
Brief Title: A Prospective/Retrospective,Randomized Controlled Clinical Study of Interferon Atomization in the 2019-nCoV Pneumonia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qin Ning, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJ20200131
Record Dates: First submitted 2020-02-02; First posted 2020-02-05 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: 2019-nCoV

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abidol hydrochloride (Experimental): Standard symptomatic support therapy (SMT) plus abidol hydrochloride(0.2g, 3 times a day).
  Interventions: Drug: Abidol hydrochloride
- Abidol Hydrochloride combined with Interferon atomization (Experimental): Interferon(PegIFN-α-2b) atomization was added(45ug, add to sterile water 2ml, twice a day) on the basis of group I.
  Interventions: Drug: Abidol Hydrochloride combined with Interferon atomization

INTERVENTIONS:
Drug: Abidol hydrochloride — 0.2g once, 3 times a day,two weeks
  Arms: Abidol hydrochloride
Drug: Abidol Hydrochloride combined with Interferon atomization — Abidol Hydrochloride:0.2g once, 3 times a day,two weeks; Interferon(PegIFN-α-2b) atomization:45ug, add to sterile water 2ml, twice a day,two weeks
  Arms: Abidol Hydrochloride combined with Interferon atomization

SUMMARY:
At present, there is no specific and effective antiviral therapy.In this study, an open, prospective/retrospective, randomized controlled cohort study was designed to compare the efficacy of two therapeutic schemes(abidol hydrochloride,abidol hydrochloride combined with interferon atomization)in the treatment of 2019-nCoV viral pneumonia, so as to provide reliable evidence-based medicine for the treatment of viral pneumonia caused by 2019-nCoV.

ELIGIBILITY:
Inclusion Criteria:

1)2019-nCoV nucleic acid test was positive. 2)CT of the lung conformed to the manifestation of viral pneumonia.

Exclusion Criteria:

1. Patients who meet any of the contraindications in the experimental drug labeling
2. Patients who do not want to participate in this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of disease remission | two weeks
  A: For mild patients : fever, cough and other symptoms relieved with improved lung CT; B:For severe patients : fever, cough and other symptoms relieved with improved lung CT,SPO2> 93% or PaO2/FiO2> 300mmHg (1mmHg=0.133Kpa);
Time for lung recovery | two weeks
  Compare the average time of lung imaging recovery after 2 weeks of treatment in each group.

SECONDARY OUTCOMES:
Rate of no fever | two weeks
Rate of respiratory symptom remission | two weeks
Rate of lung imaging recovery | two weeks
Rate of CRP,ES,Biochemical criterion (CK,ALT,Mb)recovery | two weeks
Rate of undetectable viral RNA | two weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department and Institute of Infectious Disease, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided